CLINICAL TRIAL: NCT05267431
Title: Outcomes of Different Biological Therapy on Rheumatoid Arthritis
Brief Title: Outcomes of Biological Therapy on Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nesma Mansour Mohamed, Outcomes of different biological therapy on rheumatoid arthritis, Sohag University
Other Study IDs: Soh-Med-22-02-16
Record Dates: First submitted 2022-02-14; First posted 2022-03-04 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Biological Products; Antirheumatic Agents; hydroquinone; Methotrexate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA patients recieved biological therapy: RA patients recieved different biological therapy
- RA patients recieved different DMARDS: RA patients recieved different DMARDS
  Interventions: Drug: Biological Drug

INTERVENTIONS:
Drug: Biological Drug — Different biological drugs
  Other Names: DMARDS as hydroquinone and methotrexate
  Groups: RA patients recieved different DMARDS

SUMMARY:
Evaluate effect of biological therapy on activity of RA compared to usual DMARDs

DETAILED DESCRIPTION:
Comparison between RA activity in both groups who recieved biological and DMARDS therapy

ELIGIBILITY:
Inclusion Criteria:

* RA patients

Exclusion Criteria:

* any other connective tissue disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in activity of rheumatoid arthritis | After 3 months of treatment
  By DAS 28; it include 28 tender and swollen joints, laboratory test (ESR) and visual analogue score, if it higher than 5.1 it mean high disease activity and if lower than 3.2 it mean low activity and consider remission if lower than 2.6

SECONDARY OUTCOMES:
Activity of RA | 3 months after treatment
  MHAQ.scores include questionnaire from eight activities of daily living and range from 0 to 3 and lower scores mean better function state and high scores mean worse function state

CONTACTS AND LOCATIONS:
Overall Officials: N M AHM, Specialist, Principal Investigator — Sohag faculty of medicine; M M AHM, Principal Investigator — Sohag faculty of medicine
Locations (1):
- Sohag faculty of medicine, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No